CLINICAL TRIAL: NCT06416202
Title: Comparative Efficacy of Advanced Hybrid Closed Loop (AHCL) Therapy Versus Open-Loop Insulin Delivery (OLID) System in Type 1 Diabetes Management During Ramadan: A Randomized Controlled Trial
Brief Title: Closed Loop Pumps vs. Traditional Open Loop Pumps in Managing Blood Glucose Levels in T1DM Patients Fasting in Ramadan.
Acronym: HybridRam
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Nouf Aboalsamh, Principal Investigator, King Fahad Medical City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00010471; FWA00018774 (Other: Federal Wide Assurance NlH, US)
Record Dates: First submitted 2024-04-16; First posted 2024-05-16 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Insulin Pump Therapy

STUDY DESIGN:
Intervention Model Description: A multi-center, randomized controlled trial will be conducted at King Fahad Medical City & Prince Sultan Military Medical City. The study will involve two intervention groups and one control group: one receiving open-loop insulin delivery (OLID) and the others receiving Advanced Hybrid Closed Loop (AHCL) Therapy.
  Participants will be randomly assigned to either the control group (OLID) or one of the intervention groups (AHCL). Stratified randomization will be used according to age (<18 and ≥18 years) and HbA1c (<8.5% and ≥8.5%) to avoid overrepresentation of certain age or glycemic control groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Open loop insulin delivery (Other): Patients with Type 1 Diabetes (T1D) on OLID, who observe Ramadan fasting.
  Interventions: Other: Open Loop Insulin Delivery system
- Advanced Hybrid Closed loop system (Active Comparator): AHCL system (Medtronic MiniMed 780G or Tandem T-slim x2 pump).
  Interventions: Device: Advanced hybrid closed loop insulin pump

INTERVENTIONS:
Device: Advanced hybrid closed loop insulin pump — All groups will receive comprehensive diabetes education and extensive carbohydrate counting training. Continuous glucose monitoring (CGM) will be conducted using the Guardian 4 sensor or Dexcom G6 for the intervention group depending on the type of pump used. fructosamine levels for all patients will be checked both before and after Ramadan to provide a more immediate assessment of glycemic control.
  Other Names: AHCL
  Arms: Advanced Hybrid Closed loop system
Other: Open Loop Insulin Delivery system — the control group will continue using their current CGM device. Data on glycemic control, hypoglycemic events, and patient satisfaction will be collected before and throughout Ramadan. Additionally, fructosamine levels for all patients will be checked both before and after Ramadan to provide a more immediate assessment of glycemic control.
  Other Names: OLID
  Arms: Open loop insulin delivery

SUMMARY:
Our proposed study aims to build upon the existing findings by conducting a first-of-its-kind randomized controlled trial (RCT) that directly compares Advanced Hybrid Closed Loop (AHCL) and open-loop insulin delivery (OLID) systems during Ramadan. This comparison is crucial for understanding the nuanced benefits and potential limitations of each system in the context of Ramadan fasting, a topic not yet explored in RCT settings. By undertaking this study, we intend to bridge this gap in research, providing valuable insights into the effectiveness of these contrasting insulin delivery methods. The outcomes of this research could significantly inform clinical recommendations for T1DM management during Ramadan, emphasizing the importance of personalized treatment approaches that are aligned with patient needs and technological advancements.

DETAILED DESCRIPTION:
A Multi-center, randomized controlled trial will be conducted at King Fahad Medical City and Prince Sultan Military Medical City

Participants were randomly assigned to either the control group (OLID) or one of the intervention groups (AHCL). Stratified randomization will be used according to age (<18 and ≥18 years) and HbA1c (<8.5% and ≥8.5%) to avoid overrepresentation of certain age or glycemic control groups.

All groups will receive comprehensive diabetes education and extensive carbohydrate counting training. Continuous glucose monitoring (CGM) will be conducted using the Guardian 4 sensor or Dexcom G6 for the intervention group depending on the type of pump used. The control group will continue using their current CGM device. Data on glycemic control, hypoglycemic events, and patient satisfaction will be collected before and throughout Ramadan. Additionally, fructosamine levels for all patients will be checked both before and after Ramadan to provide a more immediate assessment of glycemic control.

The investigators compared between groups in terms of the number of fasting days out of the entire month and the number of days in which participants break their fast due to diabetes-related reasons. Days when female participants do not fast due to their menstrual period will not be counted as days of fasting break for the purposes of this analysis.

Sociodemographic data, laboratory investigations, and relevant clinical data will be collected from the Electronic Health Record (EHR). CGM metrics including Time in Range (TIR), Time Above Range (TAR), Time Below Range (TBR), Glucose Management Indicator (GMI), and Coefficient of Variation (COV) will be gathered. Fructosamine levels will also be measured to assess the immediate past 2 weeks' glycemic control. A survey for diabetes distress and quality of life will be filled by the participants prior to the study.

The same CGM metrics will be collected. Insulin data including total daily dose (TDD) and percentage of basal insulin and meal boluses will be obtained. Fructosamine levels will be measured again at the end of the study to compare with the baseline measurements. This will provide a detailed assessment of the glycemic control changes specifically during Ramadan. The quality of life and diabetes distress surveys will be refilled at the end of the study. HbA1c levels will also be collected at the end of the study for a comprehensive assessment of the glycemic control during Ramadan.

Statistical Analysis:

The sample size was calculated using the confidence interval method. Statistical analyses will include comparative evaluations of HbA1c levels, hypoglycemia incidence, and patient-reported outcomes. Assuming change in time of range by 12%, power: 80% and alpha error of 5%, sample size was calculated at 25 for each group. However, we are planning to include the maximum patients we could recruit to account for the possible patients drop out.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes as per the American Diabetes Association classification for at least 1 year.
* Age 14 to 70.
* OLID therapy for at least 6 months.
* Willingness and ability to adhere to the study protocol.

Exclusion Criteria:

* Pregnancy.
* Using medications that affect blood glucose like steroids.
* Patients who are not able to fast for the entire month of Ramadan due to medical or non-medical reasons.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2025-03-29 (Estimated)

PRIMARY OUTCOMES:
Time in Range difference between AHCL and OLID during the 30 days of the month of Ramadan | 30 days (the month of Ramadan)
  Time in range on CGM (70-180mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed AlMehthel, Consultant, Principal Investigator — King Fahad Medical City
Locations (1):
- King Fahad Medical City, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wannes S, Gamal GM, Fredj MB, Al Qusayer D, El Abed S, Sedky Y, Khalil M. Glucose control during Ramadan in a pediatric cohort with type 1 diabetes on MiniMed standard and advanced hybrid closed-loop systems: A pilot study. Diabetes Res Clin Pract. 2023 Sep;203:110867. doi: 10.1016/j.diabres.2023.110867. Epub 2023 Aug 4. PMID 37544364
- [Background] Elbarbary NS, Ismail EAR. Glycemic control during Ramadan fasting in adolescents and young adults with type 1 diabetes on MiniMed 780G advanced hybrid closed-loop system: A randomized controlled trial. Diabetes Res Clin Pract. 2022 Sep;191:110045. doi: 10.1016/j.diabres.2022.110045. Epub 2022 Aug 17. PMID 35987309
- [Background] Alamoudi R, Alsubaiee M, Alqarni A, Saleh Y, Aljaser S, Salam A, Eledrisi M. Comparison of Insulin Pump Therapy and Multiple Daily Injections Insulin Regimen in Patients with Type 1 Diabetes During Ramadan Fasting. Diabetes Technol Ther. 2017 Jun;19(6):349-354. doi: 10.1089/dia.2016.0418. Epub 2017 Mar 15. PMID 28296467
- [Background] Al Awadi FF, Echtay A, Al Arouj M, Sabir Ali S, Shehadeh N, Al Shaikh A, Djaballah K, Dessapt-Baradez C, Omar Abu-Hijleh M, Bennakhi A, El Hassan Gharbi M, El Sayed El Hadidy K, Abdul Kareem Khazaal F, Hassanein MM. Patterns of Diabetes Care Among People with Type 1 Diabetes During Ramadan: An International Prospective Study (DAR-MENA T1DM). Adv Ther. 2020 Apr;37(4):1550-1563. doi: 10.1007/s12325-020-01267-4. Epub 2020 Mar 6. PMID 32144714